CLINICAL TRIAL: NCT01986400
Title: Virtual Peer-to-Peer Support Mentoring for Adolescents With Juvenile Idiopathic Arthritis: A Feasibility Pilot Randomized Controlled Trial
Brief Title: Virtual Peer-to-Peer (VP2P) Support Mentoring for Juvenile Idiopathic Arthritis (JIA): A Pilot RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Jennifer Stinson, Principal Investigator, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1000038163
Record Dates: First submitted 2013-11-11; First posted 2013-11-18 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: Adolescent; Skype; Peer Mentorship; Internet Self-Management
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Virtual Peer-to-Peer Support Mentoring (Experimental): In addition to standard medical care, adolescents in the experimental group will receive the VP2P support program, a manualized peer-mentorship program that will provide modeling and reinforcement by peers (young adults with JIA aged 16-25 years who have learned to function successfully with their JIA to the mentored participants).
  Interventions: Behavioral: Virtual Peer-to-Peer Support Mentoring
- Wait-list Control (No Intervention): The control group will receive usual care but without the mentorship intervention. They will be offered the VP2P support program after completion of outcome measures (T1 - to be completed online prior to randomization; T2 - at program completion).

INTERVENTIONS:
Behavioral: Virtual Peer-to-Peer Support Mentoring — The mentorship program will encourage mentored participants to develop and engage in self-management and transition skills and support their practice of these skills. The mentors will present information to mentored participants in a monitored virtual interaction using Skype for 8 weeks (10 total Skype sessions of 30-60 minutes each) to encourage participation in skill building tailored to their needs. All mentors will complete a paid 2.5 day training course and will be supported throughout the duration of the study (consultations with research staff to deal with unforeseen concerns). Mentored participants will complete online outcome measures prior to randomization (T1) and upon study completion (T2).
  Arms: Virtual Peer-to-Peer Support Mentoring

SUMMARY:
Study Hypothesis: A virtual peer-to-peer support intervention will improve health outcomes and quality of life in adolescents with Juvenile Idiopathic Arthritis

DETAILED DESCRIPTION:
The aim of this project is to develop and examine the impact of a virtual peer support program on health outcomes and quality of life of adolescents with Juvenile Idiopathic Arthritis using a waitlist randomized controlled trial. In addition to standard medical care, adolescents in the experimental group will receive a manualized peer mentorship program that will provide modeling and reinforcement by trained young adults aged 16-25 years who have learned to function successfully with their pain. Mentoring sessions consist of 10 sessions of 30-45 minute Skype calls over 8 weeks. Feasibility of the program will be measured in addition to quality of life, physical and emotional symptoms, pain coping, self-efficacy, social support, and self-management skills.

ELIGIBILITY:
Inclusion Criteria:

* males and females 12-18 years old
* diagnosed with Juvenile Idiopathic Arthritis (JIA) by a Rheumatologist (any sub-type)
* able to speak and read English
* access to Internet connection, computer capable of using free Skype software
* willing and able to complete online measures

Exclusion Criteria:

* significant cognitive impairments
* major co-morbid illnesses (i.e., psychiatric conditions) likely to influence HRQL assessment
* participating in peer support or self-management interventions (e.g., Teens Taking Charge).

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2013-07; Primary Completion 2015-05 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Feasibility | 2 months
  1. Accrual and Dropout Rates - recruitment and withdrawal rates will be calculated that the end of the study.
  2. Compliance (Level of Engagement) - rates of completion of weekly calls and online outcome measures will be calculated that the end of the study - defined as 100% when the participant completes 10 calls over 8 weeks with all online measures completed.
  3. Adolescents' Perception of JIA VP2P Program - the acceptability of and satisfaction with the JIA VP2P support program as measured through semi-structured phone interviews with mentees and focus groups with mentors
  4. Estimates of Intervention Effects (e.g., effect sizes, variance measures/standard deviation) on health outcomes to inform the calculation of an appropriate sample size for the future definitive multi-centred randomized controlled trial (RCT)

SECONDARY OUTCOMES:
Health-Related Quality of Life (HRQL) | Baseline, 2 months
  HRQL will be measured by using the Pediatric Quality of Life (PedsQL) Arthritis Module, a 22-item self-report scale which assesses the impact of arthritis in adolescents in terms of physical, psychological and social functioning.
Pain | Baseline, 2 months
  The Recalled Pain Inventory (RPI) measures current as well as least, average and worst pain intensity, pain unpleasantness, and pain interference with 38-items rated on a 11-point numerical rating scale (NRS).
Knowledge and Social Support | Baseline, 2 Months
  The Medical Issues, Exercise, Pain and Social Support Questionnaire (MEPS) is a 24-tem measure used to assess knowledge and social support.
Self-Efficacy | Baseline, 2 Months
  Self-efficacy is assessed using the Children's Arthritis Self-Efficacy (CASE) 11-item measure, measuring symptom management, emotional consequences and activities related to their arthritis.
Adherence | Baseline, 2 Months
  Adherence (or compliance) to prescribed medications, exercises and wearing of splints assessed using the Child Adherence Report Questionnaire (CARQ).

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer N Stinson, RN,PhD,CPNP, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Result] Stinson J, Ahola Kohut S, Forgeron P, Amaria K, Bell M, Kaufman M, Luca N, Luca S, Harris L, Victor C, Spiegel L. The iPeer2Peer Program: a pilot randomized controlled trial in adolescents with Juvenile Idiopathic Arthritis. Pediatr Rheumatol Online J. 2016 Sep 2;14(1):48. doi: 10.1186/s12969-016-0108-2. PMID 27590668
- [Result] Ahola Kohut S, Stinson J, Forgeron P, van Wyk M, Harris L, Luca S. A qualitative content analysis of peer mentoring video calls in adolescents with chronic illness. J Health Psychol. 2018 May;23(6):788-799. doi: 10.1177/1359105316669877. Epub 2016 Sep 28. PMID 27682341
- [Result] Ahola Kohut S, Stinson J, Forgeron P, Luca S, Harris L. Been There, Done That: The Experience of Acting as a Young Adult Mentor to Adolescents Living With Chronic Illness. J Pediatr Psychol. 2017 Oct 1;42(9):962-969. doi: 10.1093/jpepsy/jsx062. PMID 28340203